CLINICAL TRIAL: NCT05865249
Title: Real-world Evaluation of an Artificial-Intelligence Support Software (ArtiQ.Spiro) in Primary Care Spirometry Pathways for the Detection of Lung Disease
Brief Title: AI in PRImary Care Spirometry Pathways for Diagnosis of Lung Disease (APRIL)
Acronym: APRIL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: IRAS324175
Record Dates: First submitted 2023-04-24; First posted 2023-05-18 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Lung Diseases
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): In participants randomised to the control group, the primary care referrer will receive the spirometry report plus any additional information as per local spirometry pathway. The primary care referrer will not receive an interpretation and quality assessment report generated by ArtiQ.Spiro.
- Intervention (Other): In participants randomised to the intervention group, the primary care referrer will receive the spirometry report plus any additional information as per local spirometry pathway plus an interpretation and quality assessment report generated by ArtiQ.Spiro.
  Interventions: Other: Spirometry decision support software (ArtiQ.Spiro)

INTERVENTIONS:
Other: Spirometry decision support software (ArtiQ.Spiro) — ArtiQ.Spiro is a decision support software that combines two sub-components - one focussing on quality assessment (ArtiQ.QC), and one on spirometry interpretation (ArtiQ.PFT). It is intended to be used as an adjunct to spirometry to assist with the grading of spirometry quality and the interpretation of spirometry by providing the probability of six disease / or no disease categories.
  Other Names: ArtiQ.Spiro
  Arms: Intervention

SUMMARY:
To investigate the feasibility of performing a future real-world randomised controlled trial to determine the clinical effectiveness of ArtiQ.Spiro in supporting diagnostic performance of primary care staff in the interpretation of spirometry

DETAILED DESCRIPTION:
This is a feasibility study for a larger multicentre randomised controlled trial (RCT) assessing the impact of the ArtiQ.Spiro software on diagnostic accuracy, care processes, patient and health economic outcomes.

The primary objective of this study is to assess the feasibility of a future randomised controlled trial designed to evaluate the real-world clinical effectiveness of an artificial intelligence enabled software to support the diagnostic interpretation and quality assessment of primary care spirometry.

Endpoints of the current study will be focused on feasibility and acceptability outcomes.

Secondary objectives of this study are to collect data on potential clinical and health economic endpoints for a future randomised controlled trial designed to evaluate the real-world clinical effectiveness of an artificial intelligence enabled software to support the diagnostic interpretation and quality assessment of primary care spirometry. This will help determine the primary endpoint for a future trial and provide data to support a sample size calculation to ensure that any future trial will have adequate power.

This is a mixed methods randomised controlled feasibility trial. In PICO format:

Population: Individuals with respiratory symptoms referred clinically for primary care spirometry in Hillingdon, Leicestershire, West Hampshire.

Intervention: Local primary care spirometry pathway supported by additional artificial intelligence enabled software (ArtiQ.Spiro)

Control: Local primary care spirometry alone.

Outcomes: Feasibility outcomes with a particular focus on recruitment and retention, and acceptability of intervention and trial design. Clinical outcomes including referrer diagnostic performance and patient health status. Health economic outcomes including health care usage and economic modelling.

All participants will undergo their locally agreed spirometry pathway.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years, irrespective of sex, ethnicity, disability, sexual orientation, marital status, educational level,
* Referral by GP or nominated representative for primary care spirometry during study period.
* Patients able to provide informed consent.

Exclusion Criteria:

* Age <18yrs; Absolute contraindication to spirometry.
* Any locally defined exclusion to spirometry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2023-06-03 (Actual); Primary Completion 2024-01-22 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Identification and recruitment of eligible participants | Six months
  Contributing data: Screening & recruitment log and trial consort diagram. Progression criteria: Green (≥80% screened eligible, ≥60% eligible recruited), Amber (60-79% screened eligible, 40 - 59% eligible recruited), Red (<60% screened eligible, <40% eligible recruited)
Participant retention at follow-up | Six months
  Contributing data: Participation data and Trial Consort diagram. Progression criteria: Green (≥75% retained at 3 months, ≥60% retained at 6 months), Amber (60-75% retained at 3 months, 40-59% retained at 6 months), Red (<60% retained at 3 months, <40% retained at 6 months).
Fidelity of randomisation | Six months
  Contributing data: Numbers randomised to control/intervention groups and baseline distribution of characteristics of intervention and control groups.
  Progression criteria: Green: <10% difference in sample size, proportion of women, proportion of non-white ethnicity, proportion of > 65 years between control/intervention for each site. Amber: <15% difference in above criteria; Red: >15% difference in above criteria.
Fidelity of intervention delivery | Six months
  Contributing data: Email Logs, and Primary Care Referrer Questionnaire. Progression Criteria: Green (≥90% primary care referrers of the participants in the intervention group sent ArtiQ.Spiro report, ≥90% primary care referrers of the participants in the intervention group accessed ArtiQ.Spiro report for interpretation). Amber (85-94% primary care referrers of the participants in the intervention group sent ArtiQ.Spiro report, 75-89% primary care referrers of the participants in the intervention group accessed ArtiQ.Spiro report for interpretation). Red (<85% primary care referrers of the participants in the intervention group sent ArtiQ.Spiro report, <75% primary care referrers of the participants in the intervention group accessed ArtiQ.Spiro report for interpretation).
Contamination of control groups | Six months
  Contributing data: Email Logs. Progression Criteria: Green (≤10% primary care referrers of the participants in the control group receiving ArtiQ.Spiro report). Amber (11-15% primary care referrers of the participants in the control group receiving ArtiQ.Spiro report) Red (>15% primary care referrers of the participants in the control group receiving ArtiQ.Spiro report)
Acceptability of the intervention to referrers, spirometry practitioners and participants | Six months
  Contributing data: Stakeholder focus groups. Progression criteria: Green (Reported as acceptable (or can be with minimal modification). Amber (Reported as acceptable with modification).Red (Intervention not acceptable).
Acceptability of outcome measures and their timing | Six months
  Contributing data: Stakeholder focus groups, and Clinical Outcome Measure collection. Progression criteria: Green (Reported as acceptable or can be with minimal modification, Missing data of ≤10% for each measure).Amber (Reported as acceptable with modification, 11-25% missing data for each measure). Red: (Intervention not acceptable, >25% missing data for each measure).
Diagnostic accuracy of ArtiQ.Spiro compared with reference standard | Six months
  Contributing data: Diagnostic accuracy of ArtiQ.Spiro compared with reference standard. Progression criteria: Green: ≥ 80%, Amber: 65-79%, Red: <65%.
Data collector blinding | Six months
  Contributing data: Participation data. Progression criteria: Green (Blinding maintained for ≥85% participants), Amber (Blinding maintained for 84-70%), Red (Blinding maintained for <70%).

SECONDARY OUTCOMES:
Spirometry Quality Assessment Performance (vs Reference Standard) | Six months
  Referrers will be asked to rate the quality of the spirometry of the participant (Acceptable, usable, unusable/unacceptable) based on spirometry report (with or without ArtiQ.Spiro report). This will the be compared with Reference Standard(panel of specialists)
Primary Care Referrer Quality Assessment Confidence | Six months
  Referrers will be asked to rate the confidence in their quality assessment on a Likert scale (from 0: Very unsure to 10: Very confident).
Primary Care Referrer Technical/Pattern Interpretation | Six months
  Referrer will be asked to provide their Technical/Pattern Interpretation of the spirometry report received (Normal, Obstructive, Restrictive, Mixed), and their confidence in their technical/pattern interpretation.
Primary Care Referrer Technical/Pattern Interpretation Confidence | Six months
  Referrers will be asked to rate their confidence in their Technical/Pattern Interpretation on a Likert scale (from 0: Very unsure to 10: Very confident).
Primary Care Referrer Diagnostic Performance (versus Reference Standard) | Six months
  Referrers will be asked to provide a preferred diagnosis based on spirometry report (with/without ArtiQ.Spiro report) and information from primary care records.
Primary Care Referrer Diagnostic Confidence | Six months
  Referrers will be asked to rate the confidence in their diagnosis on a continuous visual analogue scale (from 0: Very unsure to 10: Very confident).
Patient health status | Six months
  Health Status will be measured by the EQ5D5L at baseline, 3 and 6 months post spirometry.
Heath and social care usage | Six months
  This will be measured using a Patient Healthcare Resource Use Questionnaire at baseline, 3 and 6 months post spirometry.
Health economic modelling | Six months
  The health economic analysis will compare health-related costs and benefits of ArtiQ.Spiro supported spirometry with standard spirometry pathways, as observed within the study.
Focus groups | Six months.
  Three focus groups will be conducted, comprising trial patient participants, primary care referrers and spirometry practitioners. These will be used to assess feasibility and acceptability of the trial procedures, intervention, trial outcomes.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Gillian Doe, Leicester
  - Harefield Hospital, Uxbridge

IPD SHARING:
Plan to Share IPD: No